CLINICAL TRIAL: NCT06410235
Title: The Effect of Thoracic Manipulation on Upper Body Stability in Basketball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Basketball Athletes
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic manipulation and exercise program (Experimental): Thoracic manipulation and exercise program
  Interventions: Other: Thoracic manipulation and exercise program
- exercise program (Active Comparator): exercise program
  Interventions: Other: exercise program

INTERVENTIONS:
Other: Thoracic manipulation and exercise program — The group received exercises and manipulation with physiotherapist follow-up for eight weeks and thoracic manipulation was performed once a week.
  Arms: Thoracic manipulation and exercise program
Other: exercise program — The group received exercise
  Arms: exercise program

SUMMARY:
Basketball is the most popular sport in the world and has become even more popular as a result of the attention it has received.

DETAILED DESCRIPTION:
The aim of our study was to see the effects of thoracic manipulation on upper body balance in addition to exercise programs of athletes.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals aged 14-19 years
* Being a basketball athlete
* Regular participation in training

Exclusion Criteria:

* Known neurological disorder
* Serious orthopedic conditions that prevent exercise
* Cognitive impairment

Ages: 14 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Upper Quarter Y Balance Test | 8 weeks
  A test that quantitatively analyzes an athlete's ability to reach with the free hand while maintaining weight bearing on the contralateral upper extremity. To perform the test, the athlete is asked to reach medially, inferolaterally and superolaterally with the free hand and continue weight bearing in the standard position with the standing hand.
90 Degree Push Up Test: | 8 weeks
  The 90° Push Up test is used as a measure of arm and shoulder strength and endurance. Several different forms of 90º push-up tests are used in physical fitness testing. In the past, 90º push-up tests for men were performed with toes and hands on the floor (full body push-up test).
Closed Kinetic Chain Upper Extremity Stability Test: | 8 weeks
  From the starting position they are asked to reach across their body using one hand and touch the piece of tape lying under the opposite hand. After touching the tape line, the hand returns to the original starting position. Then they do the same with the other hand. Touches are counted each time the hand reaches across the person's body and touches the tape. The total duration of the test is 15 seconds.
Polar H10: | 8 weeks
  Polar H10:is a heart rate sensor manufactured by Polar. This sensor helps athletes to accurately measure their heart rate during training.
Sorensen Test: | 8 weeks
  The lower body is secured to the table with three straps around the pelvis, knees and ankles respectively. The arms are folded across the chest while the patient is instructed to hold the upper body isometrically in a horizontal position. The time the patient holds the upper body straight and horizontal is recorded. If the test is performed for 240 seconds without problems, it is stopped.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçehir University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No